CLINICAL TRIAL: NCT02913066
Title: Prospective, Randomized, Multicenter, Phase II Noninferiority Study of S-1 Concurrent Intensity-modulated Radiation Therapy (IMRT) Versus S-1 and Cisplatin Concurrent IMRT in Inoperable Esophageal Squamous Cell Carcinoma
Brief Title: S-1 IMRT Versus S-1 and Cisplatin Concurrent IMRT in Inoperable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mianyang Central Hospital (Other)
Responsible Party: Principal Investigator, Xiaobo Du, Principal Investigator, Mianyang Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XDu
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single drug (Experimental): S-1 concurrent Radiotherapy
  Interventions: Other: S-1 concurrent radiotherapy
- Double drug (Active Comparator): S-1 plus cisplatin concurrent Radiotherapy
  Interventions: Other: S-1 plus Cisplatin concurrent radiotherapy

INTERVENTIONS:
Other: S-1 concurrent radiotherapy — Radiotherapy 60~66 Gray/28~33 times (50.4~60 Gray /28~33 planning target volume times, 60~66 Gray/28~33 Gross tumor volume of primary tumor), synchronous chemotherapy S-1 70 mg/m2 5 to 1 per week, to the end of radiotherapy. Two weeks after radiotherapy finish, two cycle adjuvant chemotherapy with S-1, 70 mg/m2, 1~ 14 days, 21 days for a cycle.
  Arms: Single drug
Other: S-1 plus Cisplatin concurrent radiotherapy — Radiotherapy 60~66 Gray/28~33 times (50.4~60 Gray /28~30 planning target volume times, Gross tumor volume of primary tumor60~66 Gray/28~33), synchronous chemotherapy S-1 70 mg/m2 1~ 14 days and 29 to 42 days, plus cisplatin 25mg/m2 1~ 4 days and 29 to 33 days. Two weeks after radiotherapy finish, two cycle adjuvant chemotherapy with S-1 70 mg/m2 1~ 14 days, plus cisplatin 25mg/m2 1~ 4 days, 21 days for a cycle.
  Arms: Double drug

SUMMARY:
Will meet the inclusion criteria of patients with esophageal squamous cell carcinoma, divided into 2 groups randomly:

Experimental group: radiotherapy combined with S-1 chemotherapy.

Control group: radiotherapy combined with S-1 chemotherapy and cisplatin.

DETAILED DESCRIPTION:
Will meet the inclusion criteria of patients with unresectable esophageal squamous cell carcinoma, divided into 2 groups randomly:

Experimental group: radiotherapy combined with S-1 chemotherapy;

control group: radiotherapy combined with S-1 chemotherapy for first to 14 days and 29 ~ 42 days, plus cisplatin first 1~ 4 days and 29 ~ 33 days. Using IMRT radiotherapy.

Two weeks after radiotherapy finish, two cycle adjuvant chemotherapy with S-1 70 mg/m2 1~ 14 days, or S-1 70 mg/m2 1~ 14 days, plus cisplatin 25mg/m2 1~ 4 days, 21 days for a cycle.

Primary Outcome Measure is complete remission rate.

Secondary Outcome Measures are overall survival (OS) and Progression-Free-Survival (PFS) and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histology or cytology confirmed esophageal squamous cell carcinoma.
2. There are measurable lesions in the RECIST standard.
3. American Joint Committee on Cancer/Union Internationale Contre le Cancer esophageal cancer staging (Sixth Edition) clinical stage II a~ IV B period.
4. Age younger than 75 years old.
5. Eastern Cooperative Oncology Group physical status score was 0 ~ 1.
6. No esophageal perforation and active esophageal bleeding, no obvious trachea, thoracic major vascular invasion.
7. Chest chemotherapy and radiotherapy, immunotherapy or biologic therapy have not been performed before.
8. Serum hemoglobin is<100g/L, platelet>100 * 109/L,Absolute neutrophil count>1.5 * 109/L.
9. Cr≤1.25 upper normal limit or CCr≥60 mL/min.
10. Serum bilirubin ≤1.5 times upper normal limit, Aspartate transaminase (SGOT) and Alanine aminotransferase (SGPT) ≤ 2.5 times upper normal limit,Alkaline phosphatase≤ 5 times upper normal limit.
11. A history of interstitial pneumonia and interstitial pneumonia.
12. FEV1>0.8 liters.
13. Patients or family members signed a formal informed consent.

Exclusion Criteria:

1. Prior to the start of the trial had received thoracic radiotherapy, chemotherapy or surgical resection of esophageal cancer.
2. Primary lesions were multifocal esophageal cancer patients, the lower bound of esophageal primary lesions was less than 3cm.
3. Patients with severe cardiovascular or pulmonary disease, interstitial pneumonia or a history of interstitial pneumonia.
4. Patients with distant metastases.
5. There were obvious esophageal ulcer, chest and back with moderate pain, and the symptoms of esophageal perforation.
6. Can't understand the test requirements, or patients may not comply with the requirements of the test.
7. There are other malignant lesion patients, but can cure skin cancer (non melanoma), cervical carcinoma in situ or malignant disease cured except for more than 5 years.
8. An allergic reaction known to have 3 or 4 levels of any treatment.
9. Had participated in other clinical trials in the past 30 days.
10. The researchers believe that some of the obvious diseases that should be excluded from this study are excluded.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate (CR) | Three months after radiotherapy finished
  Complete response rate of primary tumor which will be measured by endoscopy and computer tomography

SECONDARY OUTCOMES:
Overall Survival (OS) | Two years after adjuvant chemotherapy finished
  The time from treatment completion to patient death
Progression-Free-Survival (PFS) | Two years after adjuvant chemotherapy finished
  The time from treatment completion to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Bo Du X, Doctor, Principal Investigator — Mianyang Central Hospital
Locations (1):
- Xiaobo du, Mianyang, Sichaung, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhao Z, Wen Y, Liao D, Miao J, Gui Y, Cai H, Chen Y, Wei M, Jia Q, Tian H, Sun M, Zhang Y, Feng G, Du X. Single-Agent Versus Double-Agent Chemotherapy in Concurrent Chemoradiotherapy for Esophageal Squamous Cell Carcinoma: Prospective, Randomized, Multicenter Phase II Clinical Trial. Oncologist. 2020 Dec;25(12):e1900-e1908. doi: 10.1634/theoncologist.2020-0808. Epub 2020 Sep 28. PMID 32864805